CLINICAL TRIAL: NCT03031132
Title: The Effects of a High Protein Breakfast on Appetite and Sleep in Young Adults
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Transferring study to another University
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Heather Leidy, Associate Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2005823 HS
Record Dates: First submitted 2017-01-17; First posted 2017-01-25 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Appetite and General Nutritional Disorders
Keywords: Protein-rich breakfast; Breakfast Skipping; Young Adults; Breakfast; Food form; fMRI; Ghrelin; PYY; Sleep
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HP-Beverage Breakfast (Experimental): For 7 days, the participants will consume high protein beverage breakfast meals each morning. These meals will consist of shakes and will be 350 kcal. The macronutrient composition of these meals will contain 30 g of dietary protein, 35g CHO, and 10g fat. The HP-S and HP-B meals will be matched for energy density, sugar content, macronutrient content and types of proteins.
  Interventions: Behavioral: HP-Beverage Breakfast
- HP-Solid Breakfast (Experimental): For 7 days, the participants will consume high protein solid breakfast meals each morning. These meals will consist of traditional solid breakfast meals and will include commonly consumed breakfast foods (e.g., burritos, waffles, etc.) and will be 350 kcal. The macronutrient composition of these meals will contain 30 g of dietary protein, 35 g CHO, and 10 g fat. The HP-S and HP-B meals will be matched for energy density, sugar content, macronutrient content and types of proteins.
  Interventions: Behavioral: HP-Solid Breakfast
- Breakfast Skipping (Experimental): For 7 days, the participants will skip the morning meal. No food or calorie-containing beverages will be consumed before 12pm on acclimation days and no food consumed until ~5h post habitual breakfast time on testing day 7.
  Interventions: Behavioral: Breakfast Skipping

INTERVENTIONS:
Behavioral: HP-Beverage Breakfast — Participants will consume high protein beverage (shake) breakfast meals each morning.
  Arms: HP-Beverage Breakfast
Behavioral: HP-Solid Breakfast — Participants will consume high protein solid (traditional food items) breakfast meals each morning.
  Arms: HP-Solid Breakfast
Behavioral: Breakfast Skipping — Participants will skip breakfast each morning.
  Arms: Breakfast Skipping

SUMMARY:
The purpose of this study is to examine the effects of breakfast skipping (SKIP) vs. the consumption of a high protein solid (HP-S) breakfast vs. the consumption of a high protein beverage (HP-B) breakfast on daily appetite control, food cravings, food intake, and sleep quality in young adults.

DETAILED DESCRIPTION:
Young adults will consume the following breakfasts (in randomized order) for 7 days/pattern: 350kcal HP breakfasts (30g protein) in solid or beverage form or will skip breakfast. During the breakfast treatment periods, the participants will be provided with isocaloric breakfast meals containing 34% protein (30g protein), 40% CHO, and 26% fat. The participants will consume these meals each day throughout each of the 7 day testing periods. During the breakfast skipping treatment period, the participants will skip breakfast every morning with nothing to eat or drink (besides water) until 12:00 pm. During the acclimation days (i.e., days 1-6), participants will eat their breakfasts at home or work or simply skip the morning meal. An actigraph (to assess key indices of sleep) will be continuously worn and sleep diaries will be completed for all 7 testing days. During the afternoon of Day 3, the participant will arrive at the University of Missouri-Physical Activity and Wellness Center (MU-PAW) and fitted with a Continuous Glucose Monitor (CGM) measure glycemic control over the next 3 days. On day 6, the participant will complete hourly appetite questionnaires, consume a standardized dinner meal, and complete a salivary sample prior to sleep onset (sleep related hormones). On the 7th day of each pattern, the participants will report to the MU-PAW in the morning to complete the respective testing day. The participants will begin the testing day by either skipping breakfast or consuming their respective breakfast meal. Blood samples, salivary samples, and assessments of perceived appetite will be collected/completed at specific times throughout the day. Prior to lunch, a brain scan will be completed using functional magnetic resonance imaging (fMRI) to identify bain activation patterns in response to food pictures. Following the fMRI, the participants will be provided with an a standardized lunch. The participants will then complete the remainder of the testing day. An ad libitum food buffet will be provided for the participants to consume after their departure at home throughout the remainder of the day. . They will continue to wear the actigraph and eat/drink from the ad libitum packout cooler until going to bed that evening. Lastly, participants will complete a salivary sample and sleep diary immediately before bed. Between days 8-10, the participants will return all testing day equipment and the packout cooler, including all empty wrappers and any uneaten foods. A 3-7 day washout period will occur between patterns in which the participant will return to their habitual (i.e. pre-study) breakfast behaviors. Study outcomes include morning, mid-day, afternoon, and evening appetite, satiety, pleasure, perceived energy/sleepiness, hormonal responses (plasma glucose, insulin, ghrelin, PYY, melatonin, and cortisol concentrations), sleep indices (i.e total sleep time, sleep efficiency, perceived sleep quality), brain activation patterns, evening energy intake, and daily energy intake.

ELIGIBILITY:
Inclusion Criteria:

* age 20-32y
* BMI 22-30kg/m2
* non-smoker, non-user of tobacco products
* generally healthy (as assessed by Medical History Questionnaire)
* right-handed (fMRI requirement)
* not pregnant or lactating in the past 6 months
* not clinically diagnosed with and eating disorder
* no metabolic, hormonal, and/or neural conditions/diseases/medications that influence metabolism or food intake
* no known bleeding disorders
* not currently or previously (In the past 6 months) on a weight loss or other special diet
* no weight loss/gain (>10lbs) in the past 6 months
* normal cognitive restraint, as assessed by a score of <4 on the Three Factors Eating Habits Questionnaire (TFEQ)
* rating of ≥ 5 illustrating a minimum of "neither like nor dislike" on a 9-point hedonic scale rating for the study breakfasts
* not clinically diagnosed with obstructive sleep apnea or insomnia and does not participate in shiftwork

Exclusion Criteria:

* The potential participants will be excluded if they do not meet the inclusion criteria.

Ages: 20 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Hunger | 4 weeks
  Questionnaires, assessing appetite sensations of hunger will be completed throughout each of the testing days (which are separated by 7-10 days). The questionnaires contain validated visual analog scales (VAS) incorporating a 100 mm horizontal line rating scale for each response. The questions are worded in the following manner "how strong is your feeling of" with anchors of "not all" to "extremely."
Fullness | 4 weeks
  Questionnaires, assessing appetite sensations of fullness will be completed throughout each of the testing days (which are separated by 7-10 days). The questionnaires contain validated visual analog scales (VAS) incorporating a 100 mm horizontal line rating scale for each response. The questions are worded in the following manner "how strong is your feeling of" with anchors of "not all" to "extremely."
Prospective Food Consumption | 4 weeks
  Questionnaires, assessing appetite sensations of prospective food consumption will be completed throughout each of the testing days (which are separated by 7-10 days). The questionnaires contain validated visual analog scales (VAS) incorporating a 100 mm horizontal line rating scale for each response. The questions are worded in the following manner "how strong is your feeling of" with anchors of "not all" to "extremely."
Motivation to Eat | 4 weeks
  Questionnaires, assessing appetite sensations of motivation to eat will be completed throughout each of the testing days (which are separated by 7-10 days). The questionnaires contain validated visual analog scales (VAS) incorporating a 100 mm horizontal line rating scale for each response. The questions are worded in the following manner "how strong is your feeling of" with anchors of "not all" to "extremely."
Hedonic Ratings (pleasure) | 4 weeks
  Questionnaires, assessing appetite sensations of hedonic pleasure will be completed throughout each of the testing days (which are separated by 7-10 days). The questionnaires contain validated visual analog scales (VAS) incorporating a 100 mm horizontal line rating scale for each response. The questions are worded in the following manner "how strong is your feeling of" with anchors of "not all" to "extremely."

SECONDARY OUTCOMES:
Objective Sleep Status - Total Sleep Time | 4 weeks
  Indices of sleep status and habits will be assessed throughout the acclimation and testing days in each of the 3 study arms. The participants will wear armband accelerometers / actigraphs to measure objective sleep parameters.
Objective Sleep Quality | 4 weeks
  Indices of sleep status and habits will be assessed throughout the acclimation and testing days in each of the 3 study arms. The participants will wear armband accelerometers / actigraphs to measure objective sleep parameters.
Objective Sleep Efficiency | 4 weeks
  Indices of sleep status and habits will be assessed throughout the acclimation and testing days in each of the 3 study arms. The participants will wear armband accelerometers / actigraphs to measure objective sleep parameters.
Objective Sleep and Circadian Patterns - Salivary Cortisol | 4 weeks
  Indices of sleep status and habits salivary sampling will be completed on days 6 and 7 of each study arm to assess sleep related hormones (cortisol).
Objective Sleep and Circadian Patterns - Salivary Melatonin | 4 weeks
  Indices of sleep status and habits salivary sampling will be completed on days 6 and 7 of each study arm to assess sleep related hormones (melatonin).
Subjective Sleep Quality - Mood | 4 weeks
  Indices of perceived sleep quality (mood, energy, arousal, awakenings) will be assessed throughout the acclimation and testing days in each of the 3 study arms. The participants will complete bedtime and wake time sleep diaries to measure subjective sleep parameters.
Subjective Sleep Quality - Energy | 4 weeks
  Indices of perceived sleep quality (mood, energy, arousal, awakenings) will be assessed throughout the acclimation and testing days in each of the 3 study arms. The participants will complete bedtime and wake time sleep diaries to measure subjective sleep parameters.
Subjective Sleep Quality - Arousal | 4 weeks
  Indices of perceived sleep quality (mood, energy, arousal, awakenings) will be assessed throughout the acclimation and testing days in each of the 3 study arms. The participants will complete bedtime and wake time sleep diaries to measure subjective sleep parameters.
Subjective Sleep Quality - Awakenings | 4 weeks
  Indices of perceived sleep quality (mood, energy, arousal, awakenings) will be assessed throughout the acclimation and testing days in each of the 3 study arms. The participants will complete bedtime and wake time sleep diaries to measure subjective sleep parameters.
Functional Magnetic Resonance Imaging (fMRI) Brain Activation Responses | 4 weeks
  Brain activation responses will be assessed prior to lunch in each of the 3 testing days (separated by 2 weeks). During the fMRI brain scan procedure, the participants will focus on a set of photographs which will be projected onto a screen and easily viewed through a mirror. The fMRI paradigm incorporates stimuli from three categories of pictures including food, nonfood (animals), and blurred baseline images. Brain activation in the Insula, Amygdala, Hippocampus, and Parahippocampus will be examined when viewing food vs. animal pictures.
Evening / Dinner Energy Intake - Calories | 4 weeks
  Energy intake during dinner and evening snacks of each testing day will be measured in calories consumed.
Evening / Dinner Energy Intake - Macronutrients or food categories | 4 weeks
  Energy intake during dinner and evening snacks of each testing day will be measured as macronutrient or food category (i.e. amount of food consumed as protein, carbohydrates, fats, sugars, fiber).
Evening / Dinner Energy Intake - Food Choice | 4 weeks
  Energy intake during dinner and evening snacks of each testing day will be measured as types of foods consumed (i.e. foods typically consumed as snacks, protein-rich foods, high carbohydrate/high fat convenience foods).
Appetite and Satiety Hormones (i.e., Ghrelin, PYY) | 4 weeks
  10 total blood samples will be drawn throughout each of the testing days (which are separated by 7-10 days). Specifically, there will be seven 5 ml samples and three 9 ml samples; ~62 ml/testing day. The samples will be collected in test tubes containing EDTA (ethylenediaminetetraacetic acid). Protease inhibitors will be added to the sample to reduce protein degradation. Samples will be centrifuged at -4°C for 10 minutes. The plasma will then be separated and stored in microcentrifuge tubes at -80°C for future analysis. Appetite related hormones will be measured (ex. plasma total ghrelin and total PYY).

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Leidy, PhD, Principal Investigator — Purdue University
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Deshmukh-Taskar PR, Nicklas TA, O'Neil CE, Keast DR, Radcliffe JD, Cho S. The relationship of breakfast skipping and type of breakfast consumption with nutrient intake and weight status in children and adolescents: the National Health and Nutrition Examination Survey 1999-2006. J Am Diet Assoc. 2010 Jun;110(6):869-78. doi: 10.1016/j.jada.2010.03.023. PMID 20497776
- [Background] Nicklas TA, Yang SJ, Baranowski T, Zakeri I, Berenson G. Eating patterns and obesity in children. The Bogalusa Heart Study. Am J Prev Med. 2003 Jul;25(1):9-16. doi: 10.1016/s0749-3797(03)00098-9. PMID 12818304
- [Background] Piernas C, Popkin BM. Trends in snacking among U.S. children. Health Aff (Millwood). 2010 Mar-Apr;29(3):398-404. doi: 10.1377/hlthaff.2009.0666. PMID 20194979
- [Background] Duffey KJ, Popkin BM. Energy density, portion size, and eating occasions: contributions to increased energy intake in the United States, 1977-2006. PLoS Med. 2011 Jun;8(6):e1001050. doi: 10.1371/journal.pmed.1001050. Epub 2011 Jun 28. PMID 21738451
- [Background] Hammons AJ, Fiese BH. Is frequency of shared family meals related to the nutritional health of children and adolescents? Pediatrics. 2011 Jun;127(6):e1565-74. doi: 10.1542/peds.2010-1440. Epub 2011 May 2. PMID 21536618
- [Background] Council on Communications and Media; Strasburger VC. Children, adolescents, obesity, and the media. Pediatrics. 2011 Jul;128(1):201-8. doi: 10.1542/peds.2011-1066. Epub 2011 Jun 27. PMID 21708800
- [Background] Garcia G, Sunil TS, Hinojosa P. The fast food and obesity link: consumption patterns and severity of obesity. Obes Surg. 2012 May;22(5):810-8. doi: 10.1007/s11695-012-0601-8. PMID 22271359
- [Background] Moag-Stahlberg, A. 2010 ADAF Family nutrition and physical activity survey background data. 2010; Available from: www.Eatright.org.
- [Background] Brown AW, Bohan Brown MM, Allison DB. Belief beyond the evidence: using the proposed effect of breakfast on obesity to show 2 practices that distort scientific evidence. Am J Clin Nutr. 2013 Nov;98(5):1298-308. doi: 10.3945/ajcn.113.064410. Epub 2013 Sep 4. PMID 24004890
- [Background] Leidy HJ, Clifton PM, Astrup A, Wycherley TP, Westerterp-Plantenga MS, Luscombe-Marsh ND, Woods SC, Mattes RD. The role of protein in weight loss and maintenance. Am J Clin Nutr. 2015 Jun;101(6):1320S-1329S. doi: 10.3945/ajcn.114.084038. Epub 2015 Apr 29. PMID 25926512
- [Background] Leidy HJ, Racki EM. The addition of a protein-rich breakfast and its effects on acute appetite control and food intake in 'breakfast-skipping' adolescents. Int J Obes (Lond). 2010 Jul;34(7):1125-33. doi: 10.1038/ijo.2010.3. Epub 2010 Feb 2. PMID 20125103
- [Background] Leidy HJ, Lepping RJ, Savage CR, Harris CT. Neural responses to visual food stimuli after a normal vs. higher protein breakfast in breakfast-skipping teens: a pilot fMRI study. Obesity (Silver Spring). 2011 Oct;19(10):2019-25. doi: 10.1038/oby.2011.108. Epub 2011 May 5. PMID 21546927
- [Background] Leidy HJ, Ortinau LC, Douglas SM, Hoertel HA. Beneficial effects of a higher-protein breakfast on the appetitive, hormonal, and neural signals controlling energy intake regulation in overweight/obese, "breakfast-skipping," late-adolescent girls. Am J Clin Nutr. 2013 Apr;97(4):677-88. doi: 10.3945/ajcn.112.053116. Epub 2013 Feb 27. PMID 23446906
- [Background] Hoertel HA, Will MJ, Leidy HJ. A randomized crossover, pilot study examining the effects of a normal protein vs. high protein breakfast on food cravings and reward signals in overweight/obese "breakfast skipping", late-adolescent girls. Nutr J. 2014 Aug 6;13:80. doi: 10.1186/1475-2891-13-80. PMID 25098557
- [Background] Leidy HJ, Hoertel HA, Douglas SM, Higgins KA, Shafer RS. A high-protein breakfast prevents body fat gain, through reductions in daily intake and hunger, in "Breakfast skipping" adolescents. Obesity (Silver Spring). 2015 Sep;23(9):1761-4. doi: 10.1002/oby.21185. Epub 2015 Aug 4. PMID 26239831
- [Background] Mourao DM, Bressan J, Campbell WW, Mattes RD. Effects of food form on appetite and energy intake in lean and obese young adults. Int J Obes (Lond). 2007 Nov;31(11):1688-95. doi: 10.1038/sj.ijo.0803667. Epub 2007 Jun 19. PMID 17579632
- [Background] Leidy HJ, Bales-Voelker LI, Harris CT. A protein-rich beverage consumed as a breakfast meal leads to weaker appetitive and dietary responses v. a protein-rich solid breakfast meal in adolescents. Br J Nutr. 2011 Jul;106(1):37-41. doi: 10.1017/S0007114511000122. Epub 2011 Feb 15. PMID 21320368
- [Background] DiMeglio DP, Mattes RD. Liquid versus solid carbohydrate: effects on food intake and body weight. Int J Obes Relat Metab Disord. 2000 Jun;24(6):794-800. doi: 10.1038/sj.ijo.0801229. PMID 10878689
- [Background] Tieken SM, Leidy HJ, Stull AJ, Mattes RD, Schuster RA, Campbell WW. Effects of solid versus liquid meal-replacement products of similar energy content on hunger, satiety, and appetite-regulating hormones in older adults. Horm Metab Res. 2007 May;39(5):389-94. doi: 10.1055/s-2007-976545. PMID 17533583
- [Background] Heymsfield SB. Meal replacements and energy balance. Physiol Behav. 2010 Apr 26;100(1):90-4. doi: 10.1016/j.physbeh.2010.02.010. Epub 2010 Mar 1. PMID 20193699
- [Background] Leidy HJ, Apolzan JW, Mattes RD, Campbell WW. Food form and portion size affect postprandial appetite sensations and hormonal responses in healthy, nonobese, older adults. Obesity (Silver Spring). 2010 Feb;18(2):293-9. doi: 10.1038/oby.2009.217. Epub 2009 Jul 23. PMID 19629055
- [Background] Gwin, J. and H. Leidy, The effects of consuming high protein solid vs. beverage breakfasts on changes in body weight and body composition in overweight, breakfast skipping adolescents. The FASEB Journal, 2015. 29(1 Supplement): p. 599.1.
- [Background] Sloan, A.E., the TOP TEN Food Trends. FOOD TECHNOLOGY, 2015. 69(4): p. 24-+.
- [Background] CDC. Insufficient sleep is a public health problem. 2015 9/3/15 [cited 2016 1/15/16]; Available from: http://www.cdc.gov/features/dssleep/.
- [Background] Qin LQ, Li J, Wang Y, Wang J, Xu JY, Kaneko T. The effects of nocturnal life on endocrine circadian patterns in healthy adults. Life Sci. 2003 Sep 26;73(19):2467-75. doi: 10.1016/s0024-3205(03)00628-3. PMID 12954455
- [Background] Centers for Disease Control and Prevention (CDC). Update: West Nile virus activity--United States, 2005. MMWR Morb Mortal Wkly Rep. 2005 Sep 23;54(37):931-2. No abstract available. PMID 16180281
- [Background] Schoenborn CA, Adams PE. Health behaviors of adults: United States, 2005-2007. Vital Health Stat 10. 2010 Mar;(245):1-132. PMID 20669609
- [Background] Spiegel K, Tasali E, Penev P, Van Cauter E. Brief communication: Sleep curtailment in healthy young men is associated with decreased leptin levels, elevated ghrelin levels, and increased hunger and appetite. Ann Intern Med. 2004 Dec 7;141(11):846-50. doi: 10.7326/0003-4819-141-11-200412070-00008. PMID 15583226
- [Background] Schmid SM, Hallschmid M, Jauch-Chara K, Born J, Schultes B. A single night of sleep deprivation increases ghrelin levels and feelings of hunger in normal-weight healthy men. J Sleep Res. 2008 Sep;17(3):331-4. doi: 10.1111/j.1365-2869.2008.00662.x. Epub 2008 Jun 28. PMID 18564298
- [Background] Brondel L, Romer MA, Nougues PM, Touyarou P, Davenne D. Acute partial sleep deprivation increases food intake in healthy men. Am J Clin Nutr. 2010 Jun;91(6):1550-9. doi: 10.3945/ajcn.2009.28523. Epub 2010 Mar 31. PMID 20357041
- [Background] Benedict C, Brooks SJ, O'Daly OG, Almen MS, Morell A, Aberg K, Gingnell M, Schultes B, Hallschmid M, Broman JE, Larsson EM, Schioth HB. Acute sleep deprivation enhances the brain's response to hedonic food stimuli: an fMRI study. J Clin Endocrinol Metab. 2012 Mar;97(3):E443-7. doi: 10.1210/jc.2011-2759. Epub 2012 Jan 18. PMID 22259064
- [Background] Hogenkamp PS, Nilsson E, Nilsson VC, Chapman CD, Vogel H, Lundberg LS, Zarei S, Cedernaes J, Rangtell FH, Broman JE, Dickson SL, Brunstrom JM, Benedict C, Schioth HB. Acute sleep deprivation increases portion size and affects food choice in young men. Psychoneuroendocrinology. 2013 Sep;38(9):1668-74. doi: 10.1016/j.psyneuen.2013.01.012. Epub 2013 Feb 18. PMID 23428257
- [Background] St-Onge MP, O'Keeffe M, Roberts AL, RoyChoudhury A, Laferrere B. Short sleep duration, glucose dysregulation and hormonal regulation of appetite in men and women. Sleep. 2012 Nov 1;35(11):1503-10. doi: 10.5665/sleep.2198. PMID 23115399
- [Background] Chapman CD, Nilsson EK, Nilsson VC, Cedernaes J, Rangtell FH, Vogel H, Dickson SL, Broman JE, Hogenkamp PS, Schioth HB, Benedict C. Acute sleep deprivation increases food purchasing in men. Obesity (Silver Spring). 2013 Dec;21(12):E555-60. doi: 10.1002/oby.20579. Epub 2013 Sep 5. PMID 23908148
- [Background] Benedict C, Barclay JL, Ott V, Oster H, Hallschmid M. Acute sleep deprivation delays the glucagon-like peptide 1 peak response to breakfast in healthy men. Nutr Diabetes. 2013 Jun 24;3(6):e78. doi: 10.1038/nutd.2013.20. PMID 23797385
- [Background] Greer SM, Goldstein AN, Walker MP. The impact of sleep deprivation on food desire in the human brain. Nat Commun. 2013;4:2259. doi: 10.1038/ncomms3259. PMID 23922121
- [Background] Magee, C., et al., Acute sleep restriction alters neuroendocrine hormones and appetite in healthy male adults. Sleep and Biological Rhythms, 2009. 7: p. 125-127.
- [Background] Nedeltcheva AV, Kilkus JM, Imperial J, Kasza K, Schoeller DA, Penev PD. Sleep curtailment is accompanied by increased intake of calories from snacks. Am J Clin Nutr. 2009 Jan;89(1):126-33. doi: 10.3945/ajcn.2008.26574. Epub 2008 Dec 3. PMID 19056602
- [Background] Beebe DW, Simon S, Summer S, Hemmer S, Strotman D, Dolan LM. Dietary intake following experimentally restricted sleep in adolescents. Sleep. 2013 Jun 1;36(6):827-34. doi: 10.5665/sleep.2704. PMID 23729925
- [Background] Tanaka H, Taira K, Arakawa M, Masuda A, Yamamoto Y, Komoda Y, Kadegaru H, Shirakawa S. An examination of sleep health, lifestyle and mental health in junior high school students. Psychiatry Clin Neurosci. 2002 Jun;56(3):235-6. doi: 10.1046/j.1440-1819.2002.00997.x. PMID 12047573
- [Background] Thiagarajah, K. and M.R. Torabi, Irregular Breakfast Eating and Associated Health Behaviors: A Pilot Study among College Students. Health Educator, 2009. 41(1): p. 4-10.
- [Background] Al-Hazzaa HM, Musaiger AO, Abahussain NA, Al-Sobayel HI, Qahwaji DM. Lifestyle correlates of self-reported sleep duration among Saudi adolescents: a multicentre school-based cross-sectional study. Child Care Health Dev. 2014 Jul;40(4):533-42. doi: 10.1111/cch.12051. Epub 2013 Mar 22. PMID 23521148
- [Background] Kant AK, Graubard BI. Association of self-reported sleep duration with eating behaviors of American adults: NHANES 2005-2010. Am J Clin Nutr. 2014 Sep;100(3):938-47. doi: 10.3945/ajcn.114.085191. Epub 2014 Jul 23. PMID 25057157
- [Background] Monk TH, Reynolds CF, Kupfer DJ, Buysse DJ, Coble PA, Hayes AJ, MacHen MA, Petrie SR, Ritenour AM. The Pittsburgh Sleep Diary. J Sleep Res. 1994 Jun;3(2):111-120. PMID 10607115
- [Background] Douglas SM, Lasley TR, Leidy HJ. Consuming Beef vs. Soy Protein Has Little Effect on Appetite, Satiety, and Food Intake in Healthy Adults. J Nutr. 2015 May;145(5):1010-6. doi: 10.3945/jn.114.206987. Epub 2015 Mar 25. PMID 25809680
- [Background] Lundgren JD, Patrician TM, Breslin FJ, Martin LE, Donnelly JE, Savage CR. Evening hyperphagia and food motivation: a preliminary study of neural mechanisms. Eat Behav. 2013 Dec;14(4):447-50. doi: 10.1016/j.eatbeh.2013.08.006. Epub 2013 Aug 15. PMID 24183133
- [Derived] Gwin JA, Leidy HJ. Breakfast Consumption Augments Appetite, Eating Behavior, and Exploratory Markers of Sleep Quality Compared with Skipping Breakfast in Healthy Young Adults. Curr Dev Nutr. 2018 Aug 28;2(11):nzy074. doi: 10.1093/cdn/nzy074. eCollection 2018 Nov. PMID 30402594